CLINICAL TRIAL: NCT06500975
Title: Long Term Outcomes After Vestibular Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Labyrinth Devices, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00434328
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Bilateral Vestibular Hypofunction; Bilateral Vestibular Deficiency; Bilateral Vestibulopathy; Gentamicin Ototoxicity; Aminoglycoside Toxicity; Vestibular Diseases; Sensation Disorders; Labyrinth Diseases; Other Disorders of Vestibular Function
Keywords: Vestibular; Implant; Prosthesis; Labyrinth; Ototoxicity; Gentamicin; Oscillopsia; Disequilibrium; Dizziness; Vestibulopathy; Inner Ear
MeSH Terms: conditions — Bilateral Vestibulopathy; Vestibular Diseases; Sensation Disorders; Labyrinth Diseases; Ototoxicity; Dysequilibrium syndrome; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vestibular Implant (Experimental): Up to 32 participants will undergo implantation, activation and deactivation of a Labyrinth Devices MVI™ Multichannel Vestibular Implant System (MVI)
  Interventions: Device: Labyrinth Devices MVI™ Multichannel Vestibular Implant System

INTERVENTIONS:
Device: Labyrinth Devices MVI™ Multichannel Vestibular Implant System — Continuously motion-modulated stimulation delivered by a vestibular implant already implanted under a prior study protocol (Labyrinth Devices MVI™ Multichannel Vestibular Implant System)
  Other Names: Motion-modulated stimulation delivered by a vestibular implant already implanted under a prior study protocol

SUMMARY:
Although cochlear implants can restore hearing to individuals who have lost cochlear hair cell function, there is no widely available, adequately effective treatment for individuals suffering chronic imbalance, postural instability and unsteady vision due to bilateral vestibular hypofunction. Prior research focused on ototoxic cases has demonstrated that electrical stimulation of the vestibular nerve via a chronically implanted multichannel vestibular implant can partially restore vestibular reflexes that normally maintain steady posture and vision; improve performance on objective measures of postural stability and gait; and improve patient-reported disability and health-related quality of life. This single-arm open-label study extends that research to evaluate outcomes for up to 8 individuals with non-ototoxic bilateral vestibular hypofunction, yielding a total of fifteen adults (age 22-90 years at time of enrollment) divided as equally as possible between ototoxic and non-ototoxic cases.

DETAILED DESCRIPTION:
There is no widely available, adequately effective treatment for individuals suffering chronic imbalance, postural instability and unsteady vision due to loss of semicircular canal function despite vestibular rehabilitation exercises. The experience of 15 adults with bilateral vestibular hypofunction who underwent unilateral surgical placement of a vestibular implant and have received continuously motion-modulated electrical stimulation of the vestibular nerve for >6 months revealed vestibular implantation (VI) and motion-modulated stimulation can partially restore vestibular sensation and reflexes that normally maintain steady posture and vision. This study will examine long-term outcomes after vestibular implantation. Within constraints on power and/or minimum detectable effect size due to limits on the number of study participants permitted under IDE G150198, the study will test the following hypotheses regarding unilateral vestibular implantation, activation and long-term (≥3 years) continuous/daily use:

1. It is safe, as determined by incidence of serious unanticipated adverse device-related events and as further quantified by proportions of:

   1. implanted ears with preservation of 4-frequency pure tone average for 0.5,1,2,4 kHz air-conducted audiometric detection thresholds ≤ 50 decibel (dB) HL and ear-specific speech discrimination ≥50% (consistent with Class A or B per American Academy of Otolaryngology-Head and Neck Surgery 1995 guidelines 13 ) or ≤ 30 dB change from preoperative baseline (if preoperative baseline is ≥20 dBHL) and ear-specific speech discrimination ≤30% worse than preoperative baseline (if preoperative baseline is ≤80%)
   2. participants with preservation of useful sound-field hearing by the above criteria, and
   3. implanted ears with preservation of otolith endorgan function, if present pre-operatively
2. It is tolerable, as quantified by duration of compliance with use.
3. It is efficacious, as defined by nonzero improvement with respect to preoperative baseline gait stability as quantified by Dynamic Gait Index (DGI) and vestibulo-ocular reflex gain during passive head impulse rotation (VHITG) .

ELIGIBILITY:
Inclusion Criteria

* Adults older than 22 years old who
* have previously been enrolled in Johns Hopkins University Institutional Review Board protocol NA_00051349, IRB00335294 or IRB00346924 and
* have previously been implanted with a vestibular implant under FDA IDE G150198

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
PM1.1: Dynamic Gait Index (DGI)18 during motion-modulated implant stimulation at 4 years post-implantation, relative to pre-operative baseline, aggregated across all implant users. | 4 years post-implantation up to 5 years post-enrollment
  DGI comprises 8 gait tasks scored by an examiner: walking on a level surface, changing gait speed, walking during horizontal head turns, walking during vertical head turns, pivoting, stepping over an obstacle, stepping around obstacles, and waling up and down stairs. Each task is scored (0-3 points, 3 is best). Raw DGI score is the sum of the eight subtest scores and ranges from 0 to 24, with higher scores meaning better outcome and minimally important difference 3.2 points.
PM1.2: Gain (VHITG) of the vestibulo-ocular reflex (VOR), as measured using the video head impulse test (vHIT) | 4 years post-implantation up to 5 years post-enrollment
  During video head impulse testing (vHIT), rotational eye and head movement are measured by a goggle-mounted camera and motion sensor during brief, fast ~10 degree head rotations about the axis of a semicircular canal being tested. Performance is quantified by vestibulo-ocular reflex (VOR) gain, which a ratio of eye movement to head movement (in this case the integral of eye velocity relative to the head and the additive inverse of the integral of head velocity, respectively). VHITG, the average vHIT VOR gain for each of the three semicircular canals of the implanted ear, typically ranges from 0 to 1, with higher numbers indicating better performance.

SECONDARY OUTCOMES:
EM1.1: Vestibular Implant Composite Outcome (VICO) score | 4 years post-implantation up to 5 years post-enrollment
  Vestibular Implant Composite Outcome (VICO) score incorporates changes in vestibulo-ocular reflex gain during video head impulse testing, postural stability, gait, dizziness handicap, and health-related quality of life at 4 years post-implantation, relative to pre-operative baseline. VICO (t=6months post-op) score is the sum of changes, from preoperative baseline to 4 years post-implantation, in vestibulo-ocular reflex gain during passive head impulse rotation (VHITG); postural stability as quantified by the Bruininks-Oseretsky Test of Motor Proficiency, 2nd Edition Balance Subtest 5 (BOT); gait stability as quantified by Dynamic Gait Index (DGI); Dizziness Handicap Inventory (DHI); and SF6D health utility (SF6DU); with each component's contribution scaled to the corresponding test's minimally important difference (MID). Score 0-100, higher scores indicate better outcomes.
EM1.2: Bruininks-Oseretsky Test of Motor Proficiency 2nd Edition Balance Subtest 5 (BOT) score. | 4 years post-implantation up to 5 years post-enrollment
  BOT comprises 9 postural tasks scored by an examiner: standing with both feet on a line, standing on one leg, tandem walking, walking on a line with eyes open and eyes closed, and standing on a balance beam. Each task is performed twice and scored (0-4 points, 4 is best). The BOT score is the sum of the best scores for each task. It ranges from 0 to 36 points, with higher scores meaning better outcome and minimally important difference 4.5 points.
EM1.3: Dizziness Handicap Inventory (DHI) | 4 years post-implantation up to 5 years post-enrollment
  Dizziness Handicap Inventory (DHI) is a 25-question survey designed to quantify self-rated disability due to dizziness and unsteadiness, with scores ranging from 0 (least disabled, best outcome) to 100 (worst outcome). The minimally important difference is 18 points.
EM1.4: SF6D utility (SF6DU) score | 4 years post-implantation up to 5 years post-enrollment
  SF6DU is a unitless health utility score computed from patient-reported replies to the SF6 health-related quality of life survey and ranging from 0 to 1, with higher scores meaning better outcome and minimally important difference 0.03 points.
EM2.1: Vestibular Implant Composite Outcome (VICO) score | 4 years post-implantation up to 5 years post-enrollment
  Vestibular Implant Composite Outcome (VICO) score incorporates changes in vestibulo-ocular reflex gain during video head impulse testing, postural stability, gait, dizziness handicap, and health-related quality of life at 4 years post-implantation, relative to pre-operative baseline. VICO (t=6months post-op) score is the sum of changes, from preoperative baseline to 4 years post-implantation, in vestibulo-ocular reflex gain during passive head impulse rotation (VHITG); postural stability as quantified by the Bruininks-Oseretsky Test of Motor Proficiency, 2nd Edition Balance Subtest 5 (BOT); gait stability as quantified by Dynamic Gait Index (DGI); Dizziness Handicap Inventory (DHI); and SF6D health utility (SF6DU); with each component's contribution scaled to the corresponding test's minimally important difference (MID). Score 0-100, higher scores indicate better outcomes.
EM2.2: Bruininks-Oseretsky Test of Motor Proficiency 2nd Edition Balance Subtest 5 (BOT) | 4 years post-implantation up to 5 years post-enrollment
  BOT includes 9 postural tasks scored by an examiner: standing with both feet on a line, standing on one leg, tandem walking, walking on a line with eyes open and eyes closed, and standing on a balance beam. Each task is performed twice and scored (0-4 points). The BOT score is the sum of the best scores for each task. It ranges from 0 to 36 points, with higher scores meaning better outcome and minimally important difference 4.5 points.
EM2.3: Dizziness Handicap Inventory (DHI) | 4 years post-implantation up to 5 years post-enrollment
  Dizziness Handicap Inventory (DHI) is a 25-question survey designed to quantify self-rated disability due to dizziness and unsteadiness, with scores ranging from 0 (least disabled, best outcome) to 100 (worst outcome). The minimally important difference is 18 points.
EM2.4: SF6D utility (SF6DU) score | 4 years post-implantation up to 5 years post-enrollment
  SF6DU is a unitless health utility score computed from patient-reported replies to the SF6 health-related quality of life survey and ranging from 0 to 1, with higher scores meaning better outcome and minimally important difference 0.03 points.
EM2.5: Dynamic Gait Index (DGI) | 4 years post-implantation up to 5 years post-enrollment
  DGI comprises 8 gait tasks scored by an examiner: walking on a level surface, changing gait speed, walking during horizontal head turns, walking during vertical head turns, pivoting, stepping over an obstacle, stepping around obstacles, and waling up and down stairs. Each task is scored (0-3 points, 3 is best). Raw DGI score is the sum of the eight subtest scores and ranges from 0 to 24, with higher scores meaning better outcome and minimally important difference 3.2 points.
EM2.6: Gain (VHITG) of the vestibulo-ocular reflex (VOR), as measured using the video head impulse test (vHIT) and averaged for the three implanted semicircular canals | 4 years post-implantation up to 5 years post-enrollment
  During video head impulse testing (vHIT), rotational eye and head movement are measured by a goggle-mounted camera and motion sensor during brief, fast ~10 degree head rotations about the axis of a semicircular canal being tested. Performance is quantified by vestibulo-ocular reflex (VOR) gain, which a ratio of eye movement to head movement (in this case the integral of eye velocity relative to the head and the additive inverse of the integral of head velocity, respectively). VHITG, the average vHIT VOR gain for each of the three semicircular canals of the implanted ear, typically ranges from 0 to 1, with higher numbers indicating better performance.
EM3.1: Vestibular Implant Composite Outcome (VICO) score at 4 years post-implantation, relative to pre-operative baseline, for the subgroup of participants who have ototoxic adult-onset BVH. | 4 years post-implantation up to 5 years post-enrollment
  Vestibular Implant Composite Outcome (VICO) score incorporates changes in vestibulo-ocular reflex gain during video head impulse testing, postural stability, gait, dizziness handicap, and health-related quality of life at 4 years post-implantation, relative to pre-operative baseline. VICO (t=6months post-op) score is the sum of changes, from preoperative baseline to 4 years post-implantation, in vestibulo-ocular reflex gain during passive head impulse rotation (VHITG); postural stability as quantified by the Bruininks-Oseretsky Test of Motor Proficiency, 2nd Edition Balance Subtest 5 (BOT); gait stability as quantified by Dynamic Gait Index (DGI); Dizziness Handicap Inventory (DHI); and SF6D health utility (SF6DU); with each component's contribution scaled to the corresponding test's minimally important difference (MID). Score 0-100, higher scores indicate better outcomes.
EM3.2: Bruininks-Oseretsky Test of Motor Proficiency 2nd Edition Balance Subtest 5 (BOT) score 4 years post-implantation, relative to pre-operative baseline, for the subgroup of participants who have ototoxic adult-onset BVH. | 4 years post-implantation up to 5 years post-enrollment
  BOT includes 9 postural tasks scored by an examiner: standing with both feet on a line, standing on one leg, tandem walking, walking on a line with eyes open and eyes closed, and standing on a balance beam. Each task is performed twice and scored (0-4 points). The BOT score is the sum of the best scores for each task. It ranges from 0 to 36 points, with higher scores meaning better outcome and minimally important difference 4.5 points.
EM3.3: Dizziness Handicap Inventory (DHI) score at 4 years post-implantation, relative to pre-operative baseline, for the subgroup of participants who have ototoxic adult-onset BVH. | 4 years post-implantation up to 5 years post-enrollment
  Dizziness Handicap Inventory (DHI) is a 25-question survey designed to quantify self-rated disability due to dizziness and unsteadiness, with scores ranging from 0 (least disabled, best outcome) to 100 (worst outcome). The minimally important difference is 18 points.
EM3.4: SF6D utility (SF6DU) score at 4 years post-implantation, relative to pre-operative baseline, for the subgroup of participants who have ototoxic adult-onset BVH. | 4 years post-implantation up to 5 years post-enrollment
  SF6DU is a unitless health utility score computed from patient-reported replies to the SF6 health-related quality of life survey and ranging from 0 to 1, with higher scores meaning better outcome and minimally important difference 0.03 points.
EM3.5: Dynamic Gait Index (DGI) score at 4 years post-implantation, relative to pre-operative.baseline, for the subgroup of participants who have ototoxic adult-onset BVH. | 4 years post-implantation up to 5 years post-enrollment
  DGI comprises 8 gait tasks scored by an examiner: walking on a level surface, changing gait speed, walking during horizontal head turns, walking during vertical head turns, pivoting, stepping over an obstacle, stepping around obstacles, and waling up and down stairs. Each task is scored (0-3 points, 3 is best). Raw DGI score is the sum of the eight subtest scores and ranges from 0 to 24, with higher scores meaning better outcome and minimally important difference 3.2 points.
EM3.6: Gain (VHITG) of the vestibulo-ocular reflex, measured using the video head impulse test.averaged for the three implanted semicircular canals, relative to pre-operative baseline, for the subgroup of participants who have ototoxic adult-onset BVH. | 4 years post-implantation up to 5 years post-enrollment
  During video head impulse testing (vHIT), rotational eye and head movement are measured by a goggle-mounted camera and motion sensor during brief, fast ~10 degree head rotations about the axis of a semicircular canal being tested. Performance is quantified by vestibulo-ocular reflex (VOR) gain, which a ratio of eye movement to head movement (in this case the integral of eye velocity relative to the head and the additive inverse of the integral of head velocity, respectively). VHITG, the average vHIT VOR gain for each of the three semicircular canals of the implanted ear, typically ranges from 0 to 1, with higher numbers indicating better performance.
SM0: Type, incidence and severity of unanticipated adverse device effects as of 4 years post-implantation | 4 years post-implantation up to 5 years post-enrollment
  Assess safety of the intervention, aggregating data across all implanted participants (diversified across ototoxic and non-ototoxic/non-central adult-onset BVH), as determined by incidence of adverse device-related events from pre-intervention to 4 years post-implantation.
SM1.1: implant-side bone-conduction 4-frequency (0.5, 1, 2, 4 kHz) pure tone average detection threshold (BonePTAi) | 4 years post-implantation up to 5 years post-enrollment
  BonePTAi is the 4-frequency average of pure tone detection thresholds, in dBHL, for implant-side bone-conduction presentation of pure tones at 0.5, 1, 2 and 4 kHz. Range is -10 to 80 dBHL, with change toward smaller absolute values representing better (closer to normal) outcome.
SM1.2: implant-side air-conduction 4-frequency pure tone average detection threshold (AirPTAi) | 4 years post-implantation up to 5 years post-enrollment
  AirPTAi is the 4-frequency average of pure tone detection thresholds, in dBHL, for implant-side air-conduction presentation of pure tones at 0.5, 1, 2 and 4 kHz. Range is -10 to 120 dBHL, with change toward smaller absolute values representing better (closer to normal) outcome.
SM1.3: implant-side consonant-nucleus-consonant word discrimination score (CNCWi) | 4 years post-implantation up to 5 years post-enrollment
  CNCWi is the percentage of monosyllabic consonant-nucleus-consonant words correctly repeated when presented via an earphone speaker on the implanted side in a sound-isolation booth while a masking noise is played to the contralateral ear at 40 dB above its bone-conduction 4-frequency pure tone detection threshold if that threshold is at least 10 dB better than that of the ear being tested. CNCWi ranges from 0-100% correct, with higher score meaning better outcome.
SM1.4: sound-field Arizona Biology (AzBios)27 sentences-in-noise discrimination score | 4 years post-implantation up to 5 years post-enrollment
  AzBios is the percentage of words correctly repeated when a set of 20 Arizona Biology sentences (randomly chosen without repeats from 15 sets) is presented at a moderate level (60 dB SPL) along with masking noise (simultaneous presentation of ten sentences from another set at aggregate sound level 55 dBSPL) to both ears via a sound field speaker in a sound-isolation booth. Scores range from 0-100% correct, with higher score meaning better outcome.
SM1.5: Proportion of implanted ears that maintain American Academy of Otolaryngology - Head & Neck Surgery (AAO-HNS) 1995 Class A or B hearing13 or ≤ 30 dB change from preoperative baseline (if preoperative baseline is ≥20 dBHL) and ear-specific speech | 4 years post-implantation up to 5 years post-enrollment
  For ClassABCNCW, AAO-HNS (American Academy of Otolaryngology - Head & Neck Surgery) 1995 Class A or B hearing is defined as AirPTAi not worse than 50 dBHL and CNCWi not worse than 50%. ClassABCNCW proportion ranges from 0-100%, with higher values meaning better outcomes.
SM1.6: Proportion of implanted participants who maintain AAO-HNS 1995 Class A or B hearing or ≤ 30 dB change from preoperative baseline (if preoperative baseline is ≥20 dBHL) and ear-specific speech discrimination ≤30% worse than preoperative baseline | 4 years post-implantation up to 5 years post-enrollment
  For ClassABAzBio, AAO-HNS (American Academy of Otolaryngology - Head & Neck Surgery) 1995 Class A or B hearing is defined as AirPTAi not worse than 50 dBHL and sound-field-presentation Arizona Biology sentences-in-noise discrimination score (AzBios) not worse than 50%. ClassABAzBio proportion ranges from 0-100%, with higher values meaning better outcomes.
SM1.7: implant-side distortion-product otoacoustic emissions | 4 years post-implantation up to 5 years post-enrollment
  Distortion-product otoacoustic emissions (DPOAE) are sounds generated by a normal cochlea and detectable using a microphone in the ear canal when pairs of pure tones (centered on 0.75, 1, 1.5, 2, 3, 4, 6 and 8 kHz) are presented to the ear. DPOAE signals (and 8-valued vector for responses to stimuli centered on 0.75, 1, 1.5, 2, 3, 4, 6 and 8 kHz) are quantified in dB relative to the frequency-specific noise floor recorded by the same microphone before onset of stimulation. Response range is 0-15 dB, with higher values meaning better outcome.
SM1.8: Ear canal acoustic admittance as assessed by implant-side tympanometry | 4 years post-implantation up to 5 years post-enrollment
  Tympanometry involves using an ear canal microphone to measure ear canal acoustic admittance (conventionally reported in units of mL) and volume (in mL) by sensing reflection of a 226 Hz tone presented via a speaker in the ear canal while ear canal pressure is slowly varied from -400 to 200 decaPascals. Negative bias pressures pull the ear drum outward, positive bias pressures push the ear drum inward, and acoustic admittance is greatest when the ear drum is in a neutral anatomic position, neither retracted inward nor ballooned outward. Results are conventionally represented graphically then summarized by a three-valued vector comprising peak compliance (range 0-2 milliliters (mL), values closer to normal range of 0.3-1.4 mL meaning more normal outcome), pressure at which compliance peaks (range -400 to 200 decaPascal, values closer to 0 meaning more normal outcome), and ear canal volume (range 0-3 mL, values closer to normal adult range of 0.6-1.4 meaning more normal outcome).
SM1.9: Tinnitus Handicap Inventory (THI) | 4 years post-implantation up to 5 years post-enrollment
  The Tinnitus Handicap Inventory (THI) survey is set of questions designed to quantify self-perceived handicap due to tinnitus. THI score ranges from 0-100. Higher scores mean worse outcome.
SM1.10: Autophony Index (AI) | 4 years post-implantation up to 5 years post-enrollment
  The Autophony Index (AI) survey is set of questions designed to quantify self-perceived autophony (hearing one's voice or other internally-generated body sounds). AI score ranges from 0-104. Higher scores mean worse outcomes.
SM1.11: cervical vestibular-evoked myogenic potential (cVEMP) response amplitude | 4 years post-implantation up to 5 years post-enrollment
  Cervical vestibular-evoked myogenic potentials (cVEMPs) are a measure of saccule-mediated inhibition of sternocleidomastoid muscle electromyographic (EMG) activity during presentation of loud tones to the ipsilateral ear. After normalizing to average rectified EMG activity (in microvolts) prior to sound stimulation, cVEMP amplitudes (in microvolts) are unitless. Values range from 0 to ~10, with larger values suggesting increased saccule activity and generally indicating better outcomes, except that values above 3.0 suggest abnormally high saccule sensitivity to sound.
SM1.12: ocular vestibular-evoked myogenic potential (oVEMP) response amplitude | 4 years post-implantation up to 5 years post-enrollment
  Ocular vestibular-evoked myogenic potentials (oVEMPs) are a measure of utricle-mediated electromyographic (EMG) activity of inferior oblique and inferior rectus extraocular muscles during presentation of loud tones to the contralateral ear. Amplitude ranges from 0 to ~50 microvolts, with larger values generally suggesting increased utricle activity and better outcomes but values above 17 microvolts suggesting abnormally high utricle sensitivity to sound.
SM1.13: subjective visual vertical (SVV) as assessed using the Bucket Test | 4 years post-implantation up to 5 years post-enrollment
  A participant's vision is occluded by a bucket oriented so that its axis aligns with the participant's nasooccipital axis. The examiner rotates the bucket about the axis to a new orientation, the participant reorients it until a line drawn on the floor of the bucket is judges by the participant to be Earth-vertical and deviation of that line from true vertical is recorded. Values range over -15 to 15 degrees, with smaller absolute values meaning more normal outcomes.
SM1.14: scalp thickness at the location of implanted magnets (Tscalp) | 4 years post-implantation up to 5 years post-enrollment
  Scalp thickness at the location of implanted magnets (Tscalp) is measured in mm using a magnetic sensor. Range is 0 to 10 mm, with values closer to the range 3-7mm indicating better outcomes.
SM1.15: all adverse events, including but not limited to events related to the surgical procedure, device and device systems | 4 years post-implantation up to 5 years post-enrollment
  Assess safety of the intervention, aggregating data across all implanted participants (diversified across ototoxic and non-ototoxic/non-central adult-onset BVH), as determined by changes in hearing and otolith endorgan function indicated by changes in all adverse events, including but not limited to events related to the surgical procedure, device and device systems.
TM1: Proportion of all implanted participants who continue to use the MVI system daily at 4 years post-implantation | 4 years post-implantation up to 5 years post-enrollment
  Assess tolerance of the intervention, aggregating data across all implanted participants, as determined by the proportion of all implant recipients who continue to use the MVI system daily at 4 years post-implantation.
TM2: Proportion of implanted participants with non-ototoxic/non-central adult-onset BVH who continue to use the MVI system daily at 4 years post-implantation | 4 years post-implantation up to 5 years post-enrollment
  Assess tolerance of the intervention, for the subgroup of participants who have non-ototoxic/non-central adult-onset BVH, as determined by the proportion of implanted participants with non-ototoxic/non-central adult-onset BVH who continue to use the MVI system daily at 4 years post-implantation.
TM3: Proportion of implanted participants with ototoxic adult-onset BVH who continue to use the MVI system daily at 4 years post-implantation | 4 years post-implantation up to 5 years post-enrollment
  Assess tolerance of the intervention, for the subgroup of participants who have ototoxic adult-onset BVH, as determined by the proportion of implanted participants with ototoxic adult-onset BVH who continue to use the MVI system daily at 4 years post-implantation.

OTHER OUTCOMES:
XM1.1 (A,B,C): VOR latency during VHIT | 4 years post-implantation up to 5 years post-enrollment
  Vestibulo-ocular reflex (VOR) latency is measured in milliseconds for responses during video head impulse testing (described in 2.EM1.1) with study device providing three different modes of prosthetic vestibular nerve stimulation (A=motion-modulated/ treatment-mode stimulation, B=constant/placebo-mode stimulation, or C=no stimulation). Results are reported as a three-element vector of latencies relative to preoperative baseline (latency during mode A stimulation at 4 yr post-implantation, latency during mode B stimulation at 4 yr post-implantation, latency during mode C stimulation at 4 yr post-implantation). Latencies range from 0-1000 ms, smaller values meaning better outcome.
XM1.2 (A,B,C): saccade latency during VHIT | 4 years post-implantation up to 5 years post-enrollment
  Saccade (VOR) latency is measured in milliseconds for responses during video head impulse testing (described in 2.EM1.1) with study device providing three different modes of prosthetic vestibular nerve stimulation (A=motion-modulated/ treatment-mode stimulation, B=constant/placebo-mode stimulation, or C=no stimulation). Results are reported as a three-element vector of latencies relative to preoperative baseline (latency during mode A stimulation at 4 yr post-implantation, latency during mode B stimulation at 4 yr post-implantation, latency during mode C stimulation at 4 yr post-implantation). Latencies range from 0-1000 ms, smaller values meaning better outcome.
XM2.1 (A,B,C): VOR gain-time constant product during whole-body yaw rotary chair velocity step rotations toward the implanted ear | 4 years post-implantation up to 5 years post-enrollment
  A participant sits on a chair atop an Earth-vertical-axis rotating motor in darkness, wearing goggles that contain a camera to monitor eye rotation. The motor rotates at 240 deg/s for 1 min toward the implanted side. Slow phase nystagmus velocity is measured. Vestibulo-ocular reflex gain-time constant product GainTc is computed by multiplying gain (ratio of peak slow phase eye speed to peak chair speed) by time constant (duration after which the eye movement speed has decayed to 37% of its initial peak). GainTc ranges from 0 to 60 sec. Higher values mean better outcomes. It is measured and reported for responses during rotating chair testing with study device providing three different modes of prosthetic vestibular nerve stimulation (A=motion-modulated/ treatment-mode stimulation, B=constant/placebo-mode stimulation, or C=no stimulation). Results are reported as a 3-valued vector.
XM2.2 (A,B,C): VOR frequency response during whole-body yaw rotary chair sinusoidal rotations | 4 years post-implantation up to 5 years post-enrollment
  A participant sits on a chair atop an Earth-vertical-axis rotating motor in darkness, wearing goggles that contain a camera to monitor eye rotation. The motor rotates sinusoidally at 100 deg/s peak velocity and frequency 0.05/0.1/0.2/0.5/1 Hz. Slow phase nystagmus velocity is measured. The frequency response is a 5-element vector (one per stimulus frequency) of complex numbers, each comprising a unitless gain (eye velocity amplitude divided by chair velocity amplitude) and phase equal to 360 deg times ratio (time from peak eye velocity to peak head velocity)/(period of sinusoidal stimulus). Each gain ranges from 0 to 1; higher values mean better outcome. Each phase ranges from -180 to 180; values nearer zero mean better outcome. Frequency response is reported as a 3x5 matrix of values relative to preoperative baseline for testing with study device providing three modes of vestibular nerve stimulation: A=motion-modulated, B=constant-rate, C=off.
XM3.1: electrically-evoked vestibulo-ocular reflex (eeVOR) response peak magnitude for largest response on each electrode | 4 years post-implantation up to 5 years post-enrollment
  A participant sits on a motionless chair atop in darkness, wearing goggles that contain a camera to monitor eye rotation. The vestibular implant's stimulator delivers a series of electrical pulse trains to the inner via each electrode, one at a time. Slow phase nystagmus velocity is measured using the camera. For each canal, the largest measured nystagmus velocity is recorded. Velocities are reported as a 3-valued vector (the highest peak velocity measured for each of the three semicircular canals in the implanted ear), with values ranging from 0-300 deg/s and higher values meaning better outcomes.
XM3.2: electrically-evoked vestibulo-ocular reflex (eeVOR) response 3D misalignment for largest response on each electrode | 4 years post-implantation up to 5 years post-enrollment
  A participant sits on a motionless chair atop in darkness, wearing goggles that contain a camera to monitor eye rotation. The vestibular implant's stimulator delivers a series of electrical pulse trains to the inner via each electrode in each semicircular canal, one at a time. Slow phase nystagmus velocity is measured using the camera. For each canal, 3-dimensional (3D) misalignment (the angle in degrees between the 3D axis of peak velocity eye rotation and the 3D axis of the targeted semicircular canal) is measured for the peak nystagmus elicited by each electrode and stimulus intensity. 3D misalignment is reported as a 3-valued vector (the misalignment angles measured for each of the three semicircular canals in the implanted ear, using the electrodes and stimulus intensities that yield the largest responses approximately aligned with the target canal's axis), with values ranging from 0-180 deg and smaller values meaning better outcomes.
XM4 (A,B,C): time to failure on Modified Romberg Test with Eyes Closed on Foam | 4 years post-implantation up to 5 years post-enrollment
  The Modified Romberg Test with Eyes Closed on Foam involves having the participant stand for as long as possible on a foam pad with feet together, arms crossed, and eyes closed. Time to failure (i.e., moving out of position or opening the eyes) is measured for a maximum of 30 seconds for each of two attempts, and the longer of two measured durations is reported in seconds, with higher values meaning better outcomes. Values are measured with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/ treatment-mode, B=constant/placebo-mode, or C=no stimulation) and reported as a 3-valued vector.
XM5.1 (A,B,C): slope of change in treadmill dynamic visual acuity with increasing walking speed (LogMAR/mph) | 4 years post-implantation up to 5 years post-enrollment
  A participant's visual acuity is measured while standing still and then while walking on a treadmill at 0.5, 1, 1.5, 2, 2.5 and 3 miles per hour (mph). The slope with which visual acuity (in logarithm base 10 of the minimum angle resolved, logMAR) worsens as treadmill speed increases (in mph) is measured from a line fit to the data and reported in units of (logMAR/mph), with values ranging from 0 to -1 and less negative numbers meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/ treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM5.2 (A,B,C): maximum treadmill velocity achieved during (mph) | 4 years post-implantation up to 5 years post-enrollment
  A participant's visual acuity is measured while standing still and then while walking on a treadmill at 0.5, 1, 1.5, 2, 2.5 and 3 miles per hour (mph). The highest treadmill speed the participant tolerates is recorded in mph, with higher speeds meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM6.1 (A,B,C): gait speed when walking in well-light hall | 4 years post-implantation up to 5 years post-enrollment
  A participant walks in a well-lit hall while gait speed is measured in m/s. Speeds range from 0-2 m/s, with higher values meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM6.2 (A,B,C): gait speed when walking in dim light | 4 years post-implantation up to 5 years post-enrollment
  A participant walks in dim light while gait speed is measured in m/s. Speeds range from 0-2 m/s, with higher values meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM7.1 (A,B,C): TUG when walking in well-light hall | 4 years post-implantation up to 5 years post-enrollment
  A participant performs the Timed Up and Go (TUG) test, which comprises rising from a chair, walking to and around a pylon, then returning to the chair and sitting, in a well-lit hall. Time to complete the TUG ranges over ~5-30 seconds, with lower values meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM7.2 (A,B,C): TUG when walking in dim light | 4 years post-implantation up to 5 years post-enrollment
  A participant performs the Timed Up and Go (TUG) test, which comprises rising from a chair, walking to and around a pylon, then returning to the chair and sitting, in dim light. Time to complete the TUG ranges over ~5-30 seconds, with lower values meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM8.1 (A,B,C): gait speed when walking during dual task/cognitive distraction (Serial 7s downward counting) | 4 years post-implantation up to 5 years post-enrollment
  While counting downward in increments of -7 (from a number randomly selected between 91 and 109 by the examiner), a participant walks in a well-lit hall and gait speed is measured in m/s. Speeds range from 0-2 m/s, with higher values meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM8.2 (A,B,C): TUG during dual task/cognitive distraction (Serial 7s) | 4 years post-implantation up to 5 years post-enrollment
  While counting downward in increments of -7 (from a number randomly selected between 91 and 109 by the examiner), a participant performs the Timed Up and Go (TUG) test, which comprises rising from a chair, walking to and around a pylon, then returning to the chair and sitting, in dim light. Time to complete the TUG ranges over ~5-30 seconds, with lower values meaning better outcome. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM9 (A,B,C): Serial 7s downward counting while standing with eyes open | 4 years post-implantation up to 5 years post-enrollment
  A participant counts downward for 20 seconds in increments of -7 (from a number randomly selected between 91 and 109 by the examiner) while standing with eyes open. The number of increments correctly subtracted is counted, with higher number of increments meaning better performance. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM10.1 (A,B,C): time to complete the Trail Making Test Part B (TMT) | 4 years post-implantation up to 5 years post-enrollment
  A participant performs the Trail Making Test Part B (TMT), using a pen to connect a set of 25 pre-drawn and numbered circles on a sheet of paper as quickly as possible while being accurate. The time in seconds required to complete the test is recorded, with shorter time meaning better performance. The test is repeated with the study device providing three different modes of prosthetic stimulation (A=motion-modulated/treatment-mode, B=constant/placebo-mode, or C=no stimulation). Results are reported as a 3-valued vector.
XM10.2 (A,B,C): performance on the Triangle Completion Test (TCT) | 4 years post-implantation up to 5 years post-enrollment
  After a practice trial with eyes open, a participant performs the Triangle Completion Test (TCT). The blindfolded participant is assisted while walking slowly along 2 segments of a pre-drawn 92.5 × 185.5 × 212 cm, 30°-60°-90° triangular path and instructed to complete the final segment independently, ending at his/her best estimate of the starting point. The participant walks counterclockwise for two triangles and then clockwise for two. End point is marked midway between each foot's largest toe. Distance (in cm, range ~0-100, smaller better) from end point to starting point and angle (absolute value, range 0-180 deg, smaller better) between the participant's path and the correct path are averaged over four trials. The test is repeated with the study device providing three modes of prosthetic stimulation: A (motion-modulated), B (constant rate) and C (off). Results are reported as a 3 by 2-valued matrix.
XM11: electrode impedance | 4 years post-implantation up to 5 years post-enrollment
  Electrical impedances are measured using 26.67 microsecond/phase biphasic current pulses at 302.4 cu (clinical units) of current for each of the 9 stimulating electrodes and reported as a 9-valued vector. Values range from 0 to 25 kiloohm (kΩ). Values of <2 kΩ, abnormally low and values >15 kΩ are abnormally high, values in the range 2-15 kΩ are normal, and values closer to normal range mean better outcome. Impedances for the 9 electrodes are reported as a 9-valued vector.
XM12: electrode location distance, as determined by post-implantation computed tomography (CT) imaging | 4 years post-implantation up to 5 years post-enrollment
  For each canal, the distance between the center of crista ampullaris and the nearest stimulating electrode is measured on a post-implantation computed tomography (CT) scan in mm, with values ranging from 0-5 mm and smaller values meaning better outcome. Best-electrode distances for the 3 canals are reported as a 3-valued vector.
XM13: vestibular evoked compound action potential (veCAP)24 amplitude | 4 years post-implantation up to 5 years post-enrollment
  Peak vestibular-evoked compound action potential (veCAP) amplitude is measured for each implanted electrode and reported for the 9 implanted electrodes, with range 0-1000 microvolts and higher values meaning better outcome, as a 9-valued vector.
XM14.1: scalp thickness over the implant, measured on post-operative CT imaging | 4 years post-implantation up to 5 years post-enrollment
  Scalp thickness over the implant is measured in mm using a post-operative CT scan performed 3 weeks after implantation.
XM14.2: inductively-measured intercoil distance between implant antenna coil and external processor antenna coil | 4 years post-implantation up to 5 years post-enrollment
  Inductively-measured intercoil distance between implant antenna coil and external processor antenna coil is measured in mm 3 weeks after implantation and 4 years post-implantation, and the change between those two values is reported in mm, with numbers less than (initial thickness minus 3 mm) meaning better outcome.
XM15.1: Bilateral Vestibulopathy Questionnaire score (BVQ) | 4 years post-implantation up to 5 years post-enrollment
  The Bilateral Vestibulopathy Questionnaire English version (BVQ) is a 24-question survey intended to quantify patient-reported disease burden due to bilateral vestibular hypofunction. Each question is answered on a 6-item Likert scale, with scores for positively-worded questions reversed before scoring. After averaging scores within each of 4 construct subsets, the 4 construct values are added to yield overall BVQ score, ranging from 4 to 24. Higher score means worse outcome.
XM15.2: Number of Audio/video recording of structured interviews | 4 years post-implantation up to 5 years post-enrollment
  Audio and video recording of a participant's responses to a structure set of questions regarding symptoms of bilateral vestibular hypofunction will be made preoperatively and at 4 years postoperatively. Responses are free-format and not quantified. The number of participants who complete video/imaging will be reported.
XM16: Vestibular Activities of Daily Living score (VADL) | 4 years post-implantation up to 5 years post-enrollment
  Vestibular Activities of Daily Living (VADL) is a survey designed to quantify self-rated disability due to vestibular dysfunction. Scores range from 1 (least disabled, best outcome) to 10 (worst outcome) points.
XM17 (A,B,C): Oscillopsia Visual Analog Scale score (oVAS) | 4 years post-implantation up to 5 years post-enrollment
  The Oscillopsia Visual Analog Scale (oVAS) is a 43-question survey designed to quantify self-rated oscillopsia. Each item is answered on a 6-point Likert scale (integer scores of 0 to 5, with the score X for each negatively phrase questions transformed to 5-X before summation across all questions). Total score ranges from 0 (least oscillopsia, best outcome) to 215 (worst outcome) points.
XM18: Activities-specific Balance Confidence Scale score (ABC) | 4 years post-implantation up to 5 years post-enrollment
  The Activities-specific Balance Confidence Scale (ABC) is a 16-question survey designed to quantify self-rated confidence performing daily activities that require balance. Each item is answered on an 11-item Likert scale (from 0 to 100% confidence, in 10% increments). Total score is the average of the 16 responses and ranges from 0 (least confident, worst outcome) to 100% (most confident, best outcome).
XM19.1: Vertigo Symptom Scale score (VSS) | 4 years post-implantation up to 5 years post-enrollment
  The vertigo-balance subscale score of the Vertigo Symptom Scale is a 15-item survey designed to quantify self-rated vertigo symptom severity. Each item is answered on a 5-item Likert scale (from 0 to 4, higher meaning more frequent/worse symptoms). Total score is the sum of the 15 responses and ranges from 0 (least severe/frequent, best outcome) to 75 (worst outcome).
XM19.2: Vertigo Visual Analogue Scale score (VAS) | 4 years post-implantation up to 5 years post-enrollment
  The Vertigo Visual Analogue Scale is a 9-item visual analogue scale designed to assess the intensity of vertigo symptoms for patients in different daily situations that typically induce visual vertigo. Each item is answered on a visual analogue scale by drawing a vertical line on a 10 cm line between two anchors marked 0 and 10 (with zero (0) representing no dizziness and ten (10) representing most dizziness). Total score is the sum of the 9 responses, divided by the number of answered items, and multiplied by 10. (ranges from 0 (least severe, best outcome) to 100 (most severe, worst outcome).
XM20.1: Health Utilities Index Mark 3 (HUI) | 4 years post-implantation up to 5 years post-enrollment
  The Health Utilities Index Mark 3 is an instrument designed to measure health status and health-related quality of life. HUI Mark 3 provides a utility score ranging from 0 (worst outcome) to 1 (best outcome).
XM20.2: EuroQol 5 Dimension (EQ-5D) | 4 years post-implantation up to 5 years post-enrollment
  The EuroQOL EQ5D is a 5-dimension (mobility, self-care, usual activities, pain/discomfort, anxiety depression) instrument developed to evaluate health-related quality of life. Each of the five dimensions includes five levels of severity going from 1-5 (no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to/extreme problems (5)). Scores for each dimension are combined to obtain a total score in the form of a 5 digit code (Greater number of higher scores means worse outcome.)
XM21: Tinnitus Handicap Inventory (THI) | 4 years post-implantation up to 5 years post-enrollment
  The Tinnitus Handicap Inventory (THI) survey is set of questions designed to quantify self-perceived handicap due to tinnitus. THI score ranges from 0-100. Higher scores mean worse outcome.
XM22: Autophony Index (AI) | 4 years post-implantation up to 5 years post-enrollment
  The Autophony Index (AI) survey is set of questions designed to quantify self-perceived autophony (hearing one's voice or other internally-generated body sounds). AI score ranges from 0-104. Higher scores mean worse outcomes.
XM23.1: OTOSCOPE genetic testing panel (or equivalent panel from another Clinical Laboratory Improvement Amendments (CLIA)-certified clinical diagnostic laboratory, such as Invitae Corpl) for participants who agree to genetic testing | Preoperative baseline
  For participants with a history of nonototoxic bilateral vestibular hypofunction who agree to clinical genetic testing, a University of Iowa Molecular Otology Research Laboratory OtoSCOPE® Genetic Hearing Loss Testing v9 test will be performed on a buccal swab to determine the presence or absence of an identifiably inner ear gene abnormality, and the deidentified result will be reported.
XM23.2: Presence or absence of Mitochondrially Encoded 12S RRNA (MTRNR1) gene abnormality as assessed by genetic test panel (or equivalent) for participants with known ototoxic exposure who agree to genetic testing | Preoperative baseline
  For participants with a history of ototoxic bilateral vestibular hypofunction who agree to clinical genetic testing, an MTRNR1 genetic testing panel screen will be completed to determine the presence or absence of an MTRNR1 gene abnormality, and the deidentified result will be reported.
XM23.3: RFC1 presence or absence of an MTRNR1 gene abnormality as assessed by Ataxia/CANVAS genetic testing panel (or equivalent) for participants suspected to have CANVAS or demonstrate potential CANVAS related symptoms | Preoperative baseline
  For participants with a history of ototoxic bilateral vestibular hypofunction who agree to clinical genetic testing, an MTRNR1 genetic testing panel screen will be completed to determine the presence or absence of an MTRNR1 gene abnormality, and the deidentified result will be reported.
XM24.1: Number of intraoperative video recordings of electrode implantation | Intraoperatively
  Deidentified video of the implantation surgery will be recorded intraoperatively. The number of participants who complete intraoperative recording will be reported.
XM24.2: Number of post-implantation temporal bone CT imagings | 3 weeks post-implantation
  Deidentified images for a post-implantation temporal bone computed tomography (CT) scan will be recorded 3 weeks post-implantation. The number of participants who complete imaging will be reported.
XM25: Study visit duration (days) by activity/test/assessment | 4 years post-implantation up to 3 years post-enrollment
  Explore ways to improve efficiency of procedures for performance assessment and stimulus parameter adjustment by measuring change in study visit duration by activity/test/assessment.
XM26: Number of audio/video recording of participants' descriptions of motion percepts during eeVOR testing | 4 years post-implantation up to 3 years post-enrollment
  Deidentified audio/video of the of participants' descriptions of motion percepts during eeVOR testing. The number of participants who complete video/recording will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: John P Carey, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication of de-identified data via peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication and ending 36 months after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal and signed data access agreement. Proposals should be directed to vestibularimplant@jhmi.edu.

REFERENCES:
- [Background] Sun DQ, Lehar M, Dai C, Swarthout L, Lauer AM, Carey JP, Mitchell DE, Cullen KE, Della Santina CC. Histopathologic Changes of the Inner ear in Rhesus Monkeys After Intratympanic Gentamicin Injection and Vestibular Prosthesis Electrode Array Implantation. J Assoc Res Otolaryngol. 2015 Jun;16(3):373-87. doi: 10.1007/s10162-015-0515-y. Epub 2015 Mar 20. PMID 25790951
- [Background] Sun DQ, Ward BK, Semenov YR, Carey JP, Della Santina CC. Bilateral Vestibular Deficiency: Quality of Life and Economic Implications. JAMA Otolaryngol Head Neck Surg. 2014 Jun;140(6):527-34. doi: 10.1001/jamaoto.2014.490. PMID 24763518
- [Background] Mitchell DE, Dai C, Rahman MA, Ahn JH, Della Santina CC, Cullen KE. Head movements evoked in alert rhesus monkey by vestibular prosthesis stimulation: implications for postural and gaze stabilization. PLoS One. 2013 Oct 17;8(10):e78767. doi: 10.1371/journal.pone.0078767. eCollection 2013. PMID 24147142
- [Background] Dai C, Fridman GY, Chiang B, Rahman MA, Ahn JH, Davidovics NS, Della Santina CC. Directional plasticity rapidly improves 3D vestibulo-ocular reflex alignment in monkeys using a multichannel vestibular prosthesis. J Assoc Res Otolaryngol. 2013 Dec;14(6):863-77. doi: 10.1007/s10162-013-0413-0. Epub 2013 Sep 8. PMID 24013822
- [Background] Ward BK, Agrawal Y, Hoffman HJ, Carey JP, Della Santina CC. Prevalence and impact of bilateral vestibular hypofunction: results from the 2008 US National Health Interview Survey. JAMA Otolaryngol Head Neck Surg. 2013 Aug 1;139(8):803-10. doi: 10.1001/jamaoto.2013.3913. PMID 23949355
- [Background] Valentin NS, Hageman KN, Dai C, Della Santina CC, Fridman GY. Development of a multichannel vestibular prosthesis prototype by modification of a commercially available cochlear implant. IEEE Trans Neural Syst Rehabil Eng. 2013 Sep;21(5):830-9. doi: 10.1109/TNSRE.2013.2259261. Epub 2013 May 1. PMID 23649285
- [Background] Davidovics NS, Rahman MA, Dai C, Ahn J, Fridman GY, Della Santina CC. Multichannel vestibular prosthesis employing modulation of pulse rate and current with alignment precompensation elicits improved VOR performance in monkeys. J Assoc Res Otolaryngol. 2013 Apr;14(2):233-48. doi: 10.1007/s10162-013-0370-7. Epub 2013 Jan 26. PMID 23355001
- [Background] Fridman GY, Della Santina CC. Progress toward development of a multichannel vestibular prosthesis for treatment of bilateral vestibular deficiency. Anat Rec (Hoboken). 2012 Nov;295(11):2010-29. doi: 10.1002/ar.22581. Epub 2012 Oct 8. PMID 23044664
- [Background] Rahman MA, Dai C, Fridman GY, Davidovics NS, Chiang B, Ahn J, Hayden R, Melvin TA, Sun DQ, Hedjoudje A, Della Santina CC. Restoring the 3D vestibulo-ocular reflex via electrical stimulation: the Johns Hopkins multichannel vestibular prosthesis project. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:3142-5. doi: 10.1109/IEMBS.2011.6090857. PMID 22255006
- [Background] Dai C, Fridman GY, Davidovics NS, Chiang B, Ahn JH, Della Santina CC. Restoration of 3D vestibular sensation in rhesus monkeys using a multichannel vestibular prosthesis. Hear Res. 2011 Nov;281(1-2):74-83. doi: 10.1016/j.heares.2011.08.008. Epub 2011 Aug 26. PMID 21888961
- [Background] Dai C, Fridman GY, Chiang B, Davidovics NS, Melvin TA, Cullen KE, Della Santina CC. Cross-axis adaptation improves 3D vestibulo-ocular reflex alignment during chronic stimulation via a head-mounted multichannel vestibular prosthesis. Exp Brain Res. 2011 May;210(3-4):595-606. doi: 10.1007/s00221-011-2591-5. Epub 2011 Mar 4. PMID 21374081
- [Background] Dai C, Fridman GY, Della Santina CC. Effects of vestibular prosthesis electrode implantation and stimulation on hearing in rhesus monkeys. Hear Res. 2011 Jul;277(1-2):204-10. doi: 10.1016/j.heares.2010.12.021. Epub 2010 Dec 31. PMID 21195755
- [Background] Della Santina CC. Regaining balance with bionic ears. Sci Am. 2010 Apr;302(4):68-71. doi: 10.1038/scientificamerican0410-68. No abstract available. PMID 20349578
- [Background] Fridman GY, Davidovics NS, Dai C, Migliaccio AA, Della Santina CC. Vestibulo-ocular reflex responses to a multichannel vestibular prosthesis incorporating a 3D coordinate transformation for correction of misalignment. J Assoc Res Otolaryngol. 2010 Sep;11(3):367-81. doi: 10.1007/s10162-010-0208-5. Epub 2010 Feb 23. PMID 20177732
- [Background] Della Santina CC, Migliaccio AA, Patel AH. A multichannel semicircular canal neural prosthesis using electrical stimulation to restore 3-d vestibular sensation. IEEE Trans Biomed Eng. 2007 Jun;54(6 Pt 1):1016-30. doi: 10.1109/TBME.2007.894629. PMID 17554821
- [Background] Boutros PJ, Schoo DP, Rahman M, Valentin NS, Chow MR, Ayiotis AI, Morris BJ, Hofner A, Rascon AM, Marx A, Deas R, Fridman GY, Davidovics NS, Ward BK, Trevino C, Bowditch SP, Roberts DC, Lane KE, Gimmon Y, Schubert MC, Carey JP, Jaeger A, Della Santina CC. Continuous vestibular implant stimulation partially restores eye-stabilizing reflexes. JCI Insight. 2019 Nov 14;4(22):e128397. doi: 10.1172/jci.insight.128397. PMID 31723056
- [Background] Hedjoudje A, Schoo DP, Ward BK, Carey JP, Della Santina CC, Pearl M. Vestibular Implant Imaging. AJNR Am J Neuroradiol. 2021 Jan;42(2):370-376. doi: 10.3174/ajnr.A6991. Epub 2020 Dec 24. PMID 33361382
- [Background] Chow MR, Ayiotis AI, Schoo DP, Gimmon Y, Lane KE, Morris BJ, Rahman MA, Valentin NS, Boutros PJ, Bowditch SP, Ward BK, Sun DQ, Trevino Guajardo C, Schubert MC, Carey JP, Della Santina CC. Posture, Gait, Quality of Life, and Hearing with a Vestibular Implant. N Engl J Med. 2021 Feb 11;384(6):521-532. doi: 10.1056/NEJMoa2020457. PMID 33567192
- See also: Trial-related news updates and links to application — http://www.jhu.edu/vnel